CLINICAL TRIAL: NCT04885296
Title: Evaluation of Prototype Lenses With Experimental UV/HEV Blocker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6437
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Results first posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects will be randomized into one of two possible lens wear sequences, Test/Control.
  Interventions: Device: TRP-200; Device: JJVC Marketed Contact Lens
- Control/Test (Experimental): Eligible subjects will be randomized into one of two possible lens wear sequences, Control/Test.
  Interventions: Device: TRP-200; Device: JJVC Marketed Contact Lens

INTERVENTIONS:
Device: TRP-200 — JJVC Investigational Contact Lens
  Other Names: TEST Lens
Device: JJVC Marketed Contact Lens — ACUVUE Oasys 1-Day
  Other Names: CONTROL Lens

SUMMARY:
This is a bilateral, 2-week dispensing, randomized, controlled, subject-masked, 2×2 crossover study to evaluate the clinical performance of prototype contact lenses with experimental UV/HEV-blocker.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be between 18 and 39 (inclusive) years of age at the time of screening.
  4. By self-report, habitually wear spherical silicone hydrogel soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the past 30 days.
  5. Have a habitual contact lens prescription that is current within the prior 6 months, and they must have worn that prescription for at least 2 weeks prior to entering the study.
  6. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 through -6.00 D (except -5.00 D) in both eyes.
  7. The subject's refractive cylinder must be 1.00 D or less.
  8. The subject must have best corrected visual acuity of 20/25 or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Be currently pregnant or lactating.
  2. Have any ocular or systemic allergies or diseases that may interfere with contact lens wear.
  3. Have any autoimmune disease or use of medication, which may interfere with contact lens wear. Habitual medications used by successful soft contact lens wearers are considered acceptable.
  4. Have any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
  5. Be currently wearing lenses in a monovision, multi-focal, toric, or extended wear modality.
  6. Have participated in a contact lens or lens care product clinical trial within 14 days prior to study enrollment.
  7. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
  8. Have a history of binocular vision abnormality or strabismus.
  9. Have any infectious disease (e.g., hepatitis, tuberculosis) or contagious immunosuppressive diseases (e.g., HIV) by self-report.
  10. Have any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
  11. Have any ocular infection.
  12. Have any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
  13. Have entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or aphakia.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (12):
- United States (12):
  - Dr. James Weber & Associates, PA, Jacksonville, Florida
  - Flora Chen Poveda, OD, PA, Orange Park, Florida
  - Tallahassee Eye Center, Tallahassee, Florida
  - Visual Eyes, Roswell, Georgia
  - Birmingham Vision Care, Bloomfield Township, Michigan
  - Complete Eye Care of Medina, Medina, Minnesota
  - Dr. Debbie H. Kim, OD, Closter, New Jersey
  - Professional Vision Care, Inc., Westerville, Ohio
  - Optometry Group, LLC, Memphis, Tennessee
  - Gulf Coast Vision Center, Inc., Houston, Texas
  - Frazier Vision, Inc., Tyler, Texas
  - Botetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 228 subjects were enrolled in this study. Of those enrolled, 227 subjects were dispensed at least one study lens, while 1 subject failed to meet all eligibility criteria. Of those dispensed, 219 subjects completed the study while 8 subjects were discontinued.
Groups:
- Control (Senofilcon A C3) /Test (Senofilcon A C3): Subjects randomized to this sequence received the Control lens during the first period and Test lens during the second period.
- Test (Senofilcon A C3) /Control (Senofilcon A C3): Subjects randomized to this sequence received the Test lens during the first period and Control lens during the second period.
Period: Period 1
Arm/Group | Control (Senofilcon A C3) /Test (Senofilcon A C3) | Test (Senofilcon A C3) /Control (Senofilcon A C3)
Started | 117 | 110
Completed | 112 | 108
Not Completed | 5 | 2
Not completed — Covid-19 Related | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Test Article No Longer Available | 1 | 0
Not completed — Dispensed Study lens in Error | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Period 2
Arm/Group | Control (Senofilcon A C3) /Test (Senofilcon A C3) | Test (Senofilcon A C3) /Control (Senofilcon A C3)
Started | 112 | 108
Completed | 112 | 107
Not Completed | 0 | 1
Not completed — Subject No Longer Meets Eligibility Criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dispensed Subjects: All subjects dispensed a study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (5.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147
  Male | 80
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 19
  Black or African American | 27
  Native Hawaiian or Other Pacific Islander | 1
  White | 174
  Other | 6
Region of Enrollment [Number; unit: participants]
  United States | 227

OUTCOME MEASURES:

1. Primary Outcome: Overall Quality of Vision Score
Description: Overall quality of vision scores were assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE vision score for each lens type was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Groups:
- Test (Senofilcon A C3): Subjects that wore the Test lens in either of the two study periods.
- Control (Senofilcon A C3): Subjects that wore the Control lens in either of the two study periods.
Arm/Group | Test (Senofilcon A C3) | Control (Senofilcon A C3)
Number analyzed (Participants) | 216 | 216
Unit on a scale | 69.3 (20.84) | 69.0 (22.12)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3) vs Control (Senofilcon A C3); Test type: Non-Inferiority — Non-inferiority was declared if the lower bound of the 2-sided 95% confidence interval of the mean difference (Test - Control) was greater than -5. A 5-point increase in an average CLUE score translates into 10% shift in the distribution of scores for population of soft disposable contact lens wearers; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; LS Mean Difference = 0.4, 95% CI 2-sided [-2.2 to 3.0], Standard Error of Mean 1.32 — LS Mean difference was calculated as Test - Control

2. Secondary Outcome: Overall Comfort Scores
Description: Overall comfort scores were assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE comfort score for each lens type was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Test (Senofilcon A C3) | Control (Senofilcon A C3)
Number analyzed (Participants) | 216 | 216
Unit on a scale | 68.1 (24.58) | 69.0 (24.08)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3) vs Control (Senofilcon A C3); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; LS Mean Difference = -0.9, 95% CI 2-sided [-4.0 to 2.3], Standard Error of Mean 1.62 — LS Mean difference was calculated as Test - Control

3. Secondary Outcome: Overall Handling Scores
Description: Overall handling scores were assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE handling score for each lens type was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Test (Senofilcon A C3) | Control (Senofilcon A C3)
Number analyzed (Participants) | 216 | 216
Unit on a scale | 66.9 (23.94) | 68.6 (22.72)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3) vs Control (Senofilcon A C3); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; LS Mean Difference = -1.5, 95% CI 2-sided [-4.7 to 1.7], Standard Error of Mean 1.61 — LS Mean difference was calculated as Test - Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The study duration for each subject was approximately 26 to 30 days.
Arm/Group | Control (Senofilcon A C3) | Test (Senofilcon A C3)
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/227
Serious Adverse Events (participants affected / at risk) | 0/227 | 0/227
Other Adverse Events (participants affected / at risk) | 0/227 | 0/227

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT04885296/Prot_SAP_000.pdf